CLINICAL TRIAL: NCT05091801
Title: Effects of Increased Chewing Efficiency on the Gut Microbiome
Brief Title: Particle Size Project
Acronym: EPSOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00108805
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-09

CONDITIONS: Test if Increased Chewing Will Increased Microbiota SCFA Production
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control + Intervention (Experimental): We will explore our hypothesis using a fixed-order within-subjects study design in a group of healthy participants. Each participant will have one week of normal dietary habits and one week of increased chewing time. We will collect stool samples three times per week in order to measure microbial abundance and metabolism.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Participants will have one week of increased chewing time (chew food until they reach an apple sauce consistency)

SUMMARY:
This study is designed to test the effects of chewing efficiency on human gut microbiome composition and function.

DETAILED DESCRIPTION:
Our working hypothesis is that increased chewing will lead to an increase in short-chain fatty acid production We further expect this effect to lead to a detectable decrease in fecal particle size and distinct changes in gut microbial community composition. Here, we will explore this hypothesis using a fixed-order within-subjects study design in a group of healthy participants. Each participant will have one week of normal dietary habits and one week of increased chewing time. We will collect stool samples three times per week in order to measure microbial abundance and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Above age 18?
* Able to provide stool samples at no risk to yourself?
* Do you have card access to the CIEMAS building (work in CIEMAS, in Pratt School, or undergraduate at Duke), and are you able to visit this building (at times of your own convenience) for the purposes of this study?

Exclusion Criteria:

* Oral antibiotic treatment within the past month?
* Have a history or current diagnosis of irritable bowel syndrome?
* Have a history or current diagnosis of inflammatory bowel disease?
* Have a history or current diagnosis of type 2 diabetes?
* Have a history or current diagnosis of chronic kidney disease with decreased kidney function?
* Have a history or current diagnosis of intestinal obstruction?
* Have a history or current diagnosis of untreated colorectal cancer?
* Have you had a colonoscopy within the past month?
* Had oral antibiotics within the past month?
* Do you consume one entire non-snack meal or more per week in liquid form (smoothie, meal replacement drink, etc.)?
* Do you have any dental issues or other physical limitations that would prevent you from thoroughly chewing your food?
* Do you currently practice any mindfulness or dietary techniques that involve making sure that your food is chewed thoroughly?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
• Change in short-chain fatty acid (SCFA) measured in stool samples by gas chromatography | 1 week baseline and 1 week intervention

SECONDARY OUTCOMES:
Change in median fecal particle size as measured by laser diffraction | 1 week baseline and 1 week intervention
Change in gut microbiome composition as measured by 16S rRNA-encoding gene amplicon sequence analysis | 1 week baseline and 1 week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence David, Principal Investigator — Duke University - MGM
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No